CLINICAL TRIAL: NCT00708916
Title: Clinical and Immune-modulating Effects of CC-10004 in Discoid Lupus Erythematosus
Brief Title: Safety Study of Clinical and Immune Effects of Phosphodiesterase 4 (PDE-4) Inhibitor in Cutaneous Lupus Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-580
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Discoid Lupus Erythematosus
Keywords: Cutaneous lupus; Intervention; Discoid lupus; Phosphodiesterase 5 inhibitor
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apremilast (Experimental): CC-10004 20 mg twice daily by mouth for 12 weeks, followed by a 4 week washout period and final assessment
  Interventions: Drug: CC-10004

INTERVENTIONS:
Drug: CC-10004 — 20 mg twice daily by mouth for 12 weeks, followed by a 4 week washout period and final assessment
  Other Names: Apremilast

SUMMARY:
The purpose of this study is to determine the clinical and immunological effects of the phosphodiesterase type 4 inhibitor, CC-10004, on skin inflammation associated with cutaneous lupus erythematosus.

DETAILED DESCRIPTION:
Discoid cutaneous lupus is the most common cutaneous manifestation of lupus erythematosus, a chronic, immune mediated disease of unknown etiology. The immune processes underlying cutaneous lupus remain largely unexplored, but recent evidence suggests a role for dendritic cells (DCs), type 1 interferons (IFN) and Th1-type immune processes. Treatment of cutaneous lupus remains limited primarily to anti-malarials, with thalidomide an effective secondary agent. However, side effects associated with these treatments are potentially problematic with chronic use. Phosphodiesterases (PDE) are critical enzymes that degrade cAMP. In particular, PDE type 4 (PDE4) activity is found in inflammatory and immune cells, including DCs. The immune modulator CC-10004 is a PDE4 inhibitor with demonstrated low toxicity in phase I and II clinical studies with potential efficacy in cutaneous lupus. CC-10004 is a well-tolerated, selective PDE4 inhibitor with demonstrated inhibitory effects on Th1-type cytokines and other inflammatory mediators and is under development for the treatment of inflammatory and immune mediated conditions. Prior studies include pilot trials in psoriasis and exercise-induced asthma, with results suggesting clinical efficacy in the former study. This open label, pilot study of 16 weeks duration will explore the clinical and immune-modulating effects of CC-10004 in 10 cutaneous discoid lupus patients. Patients meeting study criteria will receive the drug for 12 weeks, followed by a 4-week washout period. Study visit time points will include weeks 0, 1, 2, 4, 6, 8, 10, 12 and 16, during which we will measure outcomes for clinical, immunological and safety parameters. To investigate early immunological changes occurring in response to treatment, we will also perform skin punch biopsies of lesional sites at week 0 and week 4 for immunohistochemical and molecular analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cutaneous discoid lupus by clinical and histopathological exam

Exclusion Criteria:

* Systemic lupus involving the internal organs
* Systemic vasculitis
* History of other clinically significant disease process
* History of HIV, hepatitis B or C
* Concurrent use of immune modulating therapy
* Evidence of incompletely treated tuberculosis
* Pregnant or lactating female

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Franks, Jr., MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Tisch Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report: PMID: 23134988 — http://jddonline.com/articles/dermatology/S1545961612P1224X — Apremilast for discoid lupus erythematosus: results of a phase 2, open-label, single-arm, pilot study. De Souza A, Strober BE, Merola JF, Oliver S, Franks AG Jr. J Drugs Dermatol. 2012 Oct;11(10):1224-6. PMID: 23134988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Drs. Franks/Oliver and other physician (attendings) would refer subjects to the unit if they were interested.
Pre-assignment Details: Screen Fail subjects were excluded from participation in trial.
Period: Overall Study
Arm/Group | Apremilast
Started | 12
Completed | 8
Not Completed | 4
Not completed — Subject Noncompliance | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Must be male or female and aged ≥ 18 years at time of consent Must have a clinical exam consistent with discoid lupus erythematosus as follows: the presence of chronic cutaneous lesions without evidence of systemic disease of lupus
Arm/Group | Apremilast
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous LE Diseases Area and Severity Index (CLASI) Score Based on Extent of Symptoms
Description: To evaluate the clinical response of cutaneous lupus patients to CC-10004. From J Invest Dermatol. 2005 Nov; 125(5): 889-894.doi: 10.1111/j.0022-202X.2005.23889.x:
  The CLASI consists of two scores. One summarizes the activity of the disease on a scale from 0 to 30, higher score translates to more severe disease. The second is a measure of the damage done by the disease on a scale form 0 to 30, higher score translates to more severe disease. Activity is scored on the basis of erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss and non-scarring alopecia. Damage is scored in terms of dyspigmentation and scarring, including scarring alopecia. Each score is reported separately. Outcome measures are reported for each time point for each subject due to the low numbers of enrollment.
Time Frame: 16 Weeks
Population: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. No study data for primary outcome measure are available
Arm/Group | Apremilast
Number analyzed (Participants) | 0

2. Secondary Outcome: Dermatology Quality of Life Index (DQLI)
Description: 1. To evaluate the clinical safety of CC-10004 in cutaneous lupus patients
  2. To determine the effect of CC-10004 on immune parameters in the skin
  3. To determine the effect of CC-10004 on immune parameters in the blood
     1. in vivo
     2. in vitro
  4. To determine the effect of CC-10004 on QOL and psychological outcome measures
Time Frame: 16 Weeks
Population: Secondary outcome measures were not measured in this study.
Arm/Group | Apremilast
Number analyzed (Participants) | 0

3. Secondary Outcome: Common Terminology Criteria for Adverse Events v3.0 (CTCAE)
Description: as for outcome 2
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 12, 16
Population: PI no longer with institution. No secondary outcome measure data available for reporting.
Arm/Group | Apremilast
Number analyzed (Participants) | 0

4. Secondary Outcome: Dermal and Circulating Blood Plasmacytoid Dendritic Cell Levels
Time Frame: Weeks 0, 4 (dermal and circulating); week 12 (circulating only)
Population: PI no longer with institution. No secondary outcome measure data available for reporting.
Arm/Group | Apremilast
Number analyzed (Participants) | 0

5. Secondary Outcome: Dermal and Circulating Blood T Regulatory Cell Levels
Description: as for outcome 2
Time Frame: Weeks 0, 4 (dermal and blood); Week 12 (blood only)
Population: PI no longer with institution. No secondary outcome measure data available for reporting.
Arm/Group | Apremilast
Number analyzed (Participants) | 0

6. Secondary Outcome: Plasma Cytokine Levels
Description: as for outcome 2
Time Frame: Weeks 0, 4, 12
Population: PI no longer with institution. No secondary outcome measure data available for reporting.
Arm/Group | Apremilast
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Apremilast
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=8)
Lichenoid Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Neuraopathy Sensory (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=8)
Nausea (Gastrointestinal disorders) | 4 (4)
Headache (Nervous system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No